CLINICAL TRIAL: NCT04444063
Title: Clinical and Radiographic Evaluation of the Non-Incised Papilla Surgical Approach With and Without Allograft Plus Platelet Rich Fibrin in Treatment of Intraosseous Defects in Stage III Periodontitis Patients: A Randomized-Controlled Clinical Trial
Brief Title: Clinical and Radiograhic Evaluation of NIPSA With and Without Allograft Plus Platelet Rich Fibrin in the Treatment of Intraosseous Defects in Stage III Periodontitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed mohamed Ibrahim Elkady, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER 3-3-3
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Periodontitis Chronic Generalized Severe; Intrabony Periodontal Defect
Keywords: minimal invasive technique; NIPSA; Allograft; PRF

STUDY DESIGN:
Intervention Model Description: it is a Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPSA technique with Allograft plus PRF (Experimental): Non-incised papilla preservation technique to treat intraosseous bony defects with the addition of Allograft plus PRF
  Interventions: Procedure: Non-Incised Papilla Surgical Approach
- NIPSA technique (Active Comparator): Non-incised papilla preservation technique to treat intraosseous bony defects without the addition of Allograft plus PRF
  Interventions: Procedure: Non-Incised Papilla Surgical Approach

INTERVENTIONS:
Procedure: Non-Incised Papilla Surgical Approach — Horizontal or oblique incision is done on the buccal mucosa as far as possible from the marginal keratinized tissue and the inter dental papilla The horizontal/oblique incision is extended mesio-distally enough to allow proper visualization of the defect A full thickness flap is elevated apico- coronally to expose the coronal limit of the defect Scaling and root planning are done using mini-curettes and power driven ultrasonic tips with care trying to maintain fibers attached to the cementum Granulation tissue is removed with mini-curettes detached from the bony walls and removed from the base of the papilla carefully with microblades and microscissors .
  1ry soft tissue closure will be performed by horizontal mattress suture 2mm from the edges of the incision as a first line of closure and then simple interrupted suture as a second line of closure using (5-0, 6-0) polypropylene suture.

SUMMARY:
Several minimal invasive techniques have been proposed since the last decade aiming to enhance and provide adequate environment for periodontal regeneration. Harrel and Rees proposed minimally invasive surgery (MIS) in 1995 and minimal invasive surgical technique (MIST) that was introduced in 2007 and then further enforced with modified minimally invasive surgical technique (M-MIST) in 2009 . A new minimal invasive technique called Non-Incised Papilla Surgical Approach (NIPSA) was introduced in 2017. It is aims to maintain the marginal tissues integrity by placing horizontal or oblique incision apical to the defect approaching the defect through apical access.

DETAILED DESCRIPTION:
Intraosseous vertical defects are one of the consequences that could result from periodontitis, which are classified according to their architecture by the number of residual walls, defect width as well as topographic extension in relation to the tooth.

Conventional surgery done for regenerative purpose regarding vertical defects has been known to be affected by clot stability, it was reported in the literature that reduced clinical outcomes occurred when early wound failure and exposure of the treated area occurred. This led to the innovation of different minimally invasive flap techniques that aimed at reducing the surgical trauma, allowing blood clot stability, protecting the regenerating site, reducing patient discomfort postoperatively as well as minimizing surgical chair time Among these techniques are papilla preservation flaps and minimally invasive surgical approaches with papilla elevation or without papilla elevation . However, these techniques had in their design incisions related to the interdental papilla which would jeopardize and complicate the vascular integrity of the interdental tissues Non incised Papilla surgical approach is a new surgical technique introduced by Moreno Rodriguez in 2017 to maintain the marginal tissues and the papilla intact by placing a horizontal or oblique incision apical to the defect and approaching it through an apical access leaving the marginal tissues to act as a "dome " protecting the blood clot

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage III periodontitis patient having at least one tooth with two wall or combined two to three walled intraosseous defect more than or equal 3 mm deep (assessed by trans-gingival probing, radiographic examination) with clinical attachment level (CAL) more than or equal 5mm and pocket depth (PD) more than or equal 6 mm.
* Defect not extending to a root furcation area.
* Vital teeth
* No history of intake of antibiotics or other medications affecting the periodontium in the previous 6 months.
* No surgical periodontal therapy carried out in the past 6 months.
* Able to sign an informed consent form.
* Patients who are cooperative, motivated, and hygiene conscious.
* Able to come for the follow up appointment's needed.

Exclusion Criteria:

* Any systemic disease that contra-indicates periodontal surgery or may affect healing.
* Smokers
* Pregnant females
* Drug abusers

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level gain (CAL) clinical attachment level gain (CAL) | 12 months
  measured with UNC periodontal probe in mm

SECONDARY OUTCOMES:
Gingival recession (GR) | 12 months
  measured with UNC periodontal probe in mm
Pocket depth (PD) | 12 months
  measured with UNC periodontal probe in mm
Radiographic defect fill | 12 months
  standardized digital periapical radiograph
Gingival bleeding | T1 T2 (Surgical phase- 8 weeks) , T4 3- months post-surgical ,T5 6-months post-surgical ,T6 1- Year post-surgical
  Gingival bleeding score
Plaque index | 12 months
  Plaque Index score
Post-surgical patient Satisfaction | 12 months
  (1-7) point scale

CONTACTS AND LOCATIONS:
Overall Officials: Omneya Abo-Eldahab, PHD, Study Chair — Cairo University; Omneya K. Tawfeek, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
I will check with my study chairs

REFERENCES:
- [Background] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Supra-alveolar attachment gain in the treatment of combined intra-suprabony periodontal defects by non-incised papillae surgical approach. J Clin Periodontol. 2019 Sep;46(9):927-936. doi: 10.1111/jcpe.13158. Epub 2019 Jul 22. PMID 31190409